CLINICAL TRIAL: NCT03478800
Title: The Feasibility and Effects of Acupuncture on Muscle Soreness and Sense of Well-being in an Adolescent Football Population.
Brief Title: Acupuncture in Adolescent Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Edward R. Laskowski, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-003475
Record Dates: First submitted 2017-06-15; First posted 2018-03-27 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Acupuncture Therapy; Sports Medicine
MeSH Terms: interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High school football players and acupuncture (Experimental): 50 healthy high school football players without active musculoskeletal injury
  Interventions: Procedure: Acupuncture

INTERVENTIONS:
Procedure: Acupuncture — Each treatment would take approximately 15-20 minutes and would take place immediately after practice for a total of five treatments. The needles are standard (0.2mm diameter #36 gauge 1 inch stainless steel) and during each treatment, 3-6 needles would be placed in the lower extremity in any of the following muscle groups: quadriceps, hamstrings, anterior tibialis, gastrocnemius-soleus complex, medial head of the gastrocnemius, peroneal muscles, or iliotibial band. The athletes would complete brief pre- and post-treatment surveys.

SUMMARY:
Is it feasible to perform acupuncture in the training field after sport performance in adolescent football players?

Does acupuncture provide a decrease in muscle soreness and improvement in overall sense of well-being in the adolescent football population?

DETAILED DESCRIPTION:
Previous studies on the effects of acupuncture on performance and post-exercise recovery have shown that it reduces perceived pain arising from exercise induced muscle soreness and reduces muscle spasm. Acupuncture has also been shown to serve as an adjunct to improve muscle strength training and to accelerate recovery from workouts and injury.

The investigators' goal is to study approximately 50 high school football players in their true pre-season warm weather training environment. The investigators will measure the effects of acupuncture treatment on muscle soreness and overall sense of well-being by administering pre- and post-treatment surveys. Athletes will undergo five treatment sessions over the course of 2.5 weeks. The treatments will be performed by licensed acupuncturists employed at Mayo Clinic. The study has been approved by the Institutional Review Board at the Mayo Clinic.

ELIGIBILITY:
Inclusion Criteria

1. Male or female members of the two local high school football teams
2. Age 13-18 years
3. No current musculoskeletal injuries
4. Generally healthy individuals who plan to complete the season barring injury or other unexpected events.

Exclusion Criteria:

1. Acupuncture treatment within the past year
2. Known active musculoskeletal injury or condition, immunocompromised state, prosthetic heart valve, pregnancy or known history of bleeding disorder.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Change in muscle soreness after post-exercise acupuncture therapy | immediately before and after acupuncture during the study period (2.5 weeks)
  Musculoskeletal pain or soreness will be measured by a Football Acupuncture Survey designed by the investigators. Participants will first be asked if they had muscle soreness or pain in the last 24-48 hours and if so, if they used any modalities to alleviate it (ice, heat, massage etc) or medications (and if so, which ones). Participants will then be asked about the presence and location of current muscle soreness and to rate the soreness on a 10 point scale with 0 being 'no muscle soreness' and 10 being 'muscle soreness as bad as can be. After acupuncture treatment, they will be the same question. The investigators will evaluate the difference between pre- and post-treatment muscle soreness.

SECONDARY OUTCOMES:
Sense of well-being | immediately before and after acupuncture, during the study period (2.5 weeks)
  'Sense of well-being' will be measured by a Football Acupuncture Survey designed by the investigators. Sense of well-being is defined on the survey as 'feeling content, happy, healthy, full of energy or relaxed while not feeling upset, anxious or fatigued.' Participants will be asked to rate their overall sense of well-being on a 10 point scale with 0 being 'as bad as it can be' and 10 being 'as good as it can be.' After acupuncture treatment, they will be the same question. The investigators will evaluate the difference between pre- and post-treatment sense of well-being.

OTHER OUTCOMES:
Presence or absence of side effects from acupuncture treatment | immediately before and after acupuncture, during the study period (2.5 weeks)
  As part of the Survey, after each treatment, participants will also be asked if they experienced side effects from the treatment that day, including but not limited to acupuncture site pain, numbness, tingling, sensations of cold or heat, and dizziness.
Overall experience and willingness to recommend or consider acupuncture in the future. | immediately before and after acupuncture, during the study period (2.5 weeks)
  As part of the Survey, participants will be asked to rate their overall experience after acupuncture after the treatment that day (poor, fair, good, very good, and excellent); whether or not they would recommend acupuncture to other teammates or athletes (yes/no); and whether or not they would consider acupuncture in the future (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Edward R Laskowski, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luetmer MT, Do A, Canzanello NC, Bauer BA, Laskowski ER. The Feasibility and Effects of Acupuncture on Muscle Soreness and Sense of Well-being in an Adolescent Football Population. Am J Phys Med Rehabil. 2019 Nov;98(11):964-970. doi: 10.1097/PHM.0000000000001226. PMID 31135462